CLINICAL TRIAL: NCT06112379
Title: A Phase III, Open-label, Randomised Study of Neoadjuvant Datopotamab Deruxtecan (Dato-DXd) Plus Durvalumab Followed by Adjuvant Durvalumab With or Without Chemotherapy Versus Neoadjuvant Pembrolizumab Plus Chemotherapy Followed by Adjuvant Pembrolizumab With or Without Chemotherapy for the Treatment of Adult Patients With Previously Untreated Triple-Negative or Hormone Receptor-low/HER2-negative Breast Cancer (D926QC00001; TROPION-Breast04)
Brief Title: A Phase III Randomised Study to Evaluate Dato-DXd and Durvalumab for Neoadjuvant/Adjuvant Treatment of Triple-Negative or Hormone Receptor-low/HER2-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D926QC00001; 2023-505928-59-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-12; First posted 2023-11-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer;; Dato-DXd; DS1062a;; TROP2;; TNBC;; HR low:; Datopotamab deruxtecan;; Antibody Drug Conjugate;; ADC;; neoadjuvant therapy;; adjuvant therapy;; durvalumab;; PD-L1;; immune-checkpoint inhibitor (ICI);
MeSH Terms: conditions — Breast Neoplasms | interventions — durvalumab; pembrolizumab; Doxorubicin; Epirubicin; Cyclophosphamide; Paclitaxel; Carboplatin; Capecitabine; olaparib

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 ratio to one of two intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dato-DXd plus durvalumab (Experimental): Participants receive durvalumab every 3 weeks (Q3W) + Dato-DXd Q3W as neoadjuvant therapy prior to surgery; followed by 9 cycles of durvaluamb Q3W as adjuvant therapy post-surgery. Adjuvant chemotherapy may be given in combination with durvalumab only if participants have residual disease.
  Olaparib may be given for participants with gBRCA-positive tumours and residual disease
  Adjuvant chemotherapy may be one of these:
  1. Doxorubicin (Q3W) or epirubicin (Q3W) + cyclophosphamide (Q3W) for 4 cycles (12 weeks) followed by paclitaxel (weekly) and carboplatin (weekly or Q3W) for 4 cycles (12 weeks);
  2. Doxorubicin (Q3W) or epirubicin (Q3W) + cyclophosphamide (Q3W) for 4 cycles (12 weeks) followed by paclitaxel (weekly) for 4 cycles (12 weeks);
  3. Carboplatin (weekly or Q3W) + paclitaxel (weekly) for 4 cycles (12 weeks);
  4. Capecitabine (Q3W) for 8 cycles.
  Interventions: Drug: Dato-DXd; Drug: Durvalumab; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin; Drug: Capecitabine; Drug: Olaparib
- Pembrolizumab plus chemotherapy (Active Comparator): Participants receive pembrolizumab every 3 weeks (Q3W) + paclitaxel weekly + carboplatin (weekly or Q3W) x 4 cycles, followed by pembrolizumab Q3W + (doxorubicin OR epirubicin) + cyclophosphamide Q3W x 4 cycles as neoadjuvant therapy prior to surgery; followed by 9 cycles of pembrolizumab Q3W as adjuvant therapy post-surgery. Adjuvant capecitabine (Q3W) for 8 cycles may be given in combination with pembrolizumab only if participants have residual disease. Olaparib may be given for participants with gBRCA-positive tumours and residual disease.
  Interventions: Drug: Pembrolizumab; Drug: Doxorubicin; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Drug: Carboplatin; Drug: Capecitabine; Drug: Olaparib

INTERVENTIONS:
Drug: Dato-DXd — Experimental drug IV infusion
  Other Names: Datopotamab deruxtecan (Dato-DXd, DS-1062a)
  Arms: Dato-DXd plus durvalumab
Drug: Durvalumab — Experimental drug IV Infusion
  Other Names: MEDI4736
  Arms: Dato-DXd plus durvalumab
Drug: Pembrolizumab — IV Infusion Active comparator
  Other Names: KEYTRUDA®
  Arms: Pembrolizumab plus chemotherapy
Drug: Doxorubicin — IV infusion Experimental/Active Comparator
Drug: Epirubicin — IV Infusion Experimental/Active Comparator
Drug: Cyclophosphamide — IV infusion Experimental/Active Comparator
Drug: Paclitaxel — IV infusion Experimental/Active Comparator
Drug: Carboplatin — IV infusion Experimental/Active Comparator
Drug: Capecitabine — Tablet Oral route of administration Experimental/Active Comparator
  Other Names: XELODA®, Capecitabine Cell Pharm, Capecitabine EG, Capecitabine Accord
Drug: Olaparib — Tablet Oral route of administration Experimental/Active Comparator
  Other Names: LYNPARZA®

SUMMARY:
This is a Phase III, 2-arm, randomised, open-label, multicentre, global study assessing the efficacy and safety of neoadjuvant Dato-DXd plus durvalumab followed by adjuvant durvalumab with or without chemotherapy compared with neoadjuvant pembrolizumab plus chemotherapy followed by adjuvant pembrolizumab with or without chemotherapy in participants with previously untreated TNBC or hormone receptor-low/HER2-negative breast cancer.

DETAILED DESCRIPTION:
The primary objectives of the study are to demonstrate superiority of neoadjuvant Dato-DXd plus durvalumab followed by adjuvant durvalumab with or without chemotherapy relative to neoadjuvant pembrolizumab plus chemotherapy followed by adjuvant pembrolizumab with or without chemotherapy in participants with previously untreated TNBC or hormone receptor-low/HER2-negative breast cancer, by investigator assessment of EFS.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years, at the time of signing the ICF.
* Histologically confirmed Stage II or III unilateral or bilateral primary invasive TNBC or hormone receptor-low/HER2-negative breast cancer
* ECOG PS of 0 or 1
* Provision of acceptable tumor sample
* Adequate bone marrow reserve and organ function
* Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies and aligned with protocol requirements.

Exclusion criteria:

* History of any prior invasive breast malignancy
* History of another primary malignancy except for malignancy treated with curative intent with no known active disease within 5 years before randomization.
* active or prior documented autoimmune or inflammatory disorders.
* Evidence of distant disease.
* Clinically significant corneal disease.
* Has active or uncontrolled hepatitis B or C virus infection.
* Known HIV infection that is not well controlled.
* Uncontrolled infection requiring i.v. antibiotics, antivirals or antifungals; suspected infections; or inability to rule out infections.
* Known to have active tuberculosis infection
* Mean resting corrected QTcF interval > 470 ms obtained from ECG
* Uncontrolled or significant cardiac disease.
* History of non-infectious ILD/pneumonitis
* Has severe pulmonary function compromise
* Any prior or concurrent surgery, radiotherapy or systemic anticancer therapy for TNBC or hormone receptor-low/HER2-negative breast cancer
* For females only: is pregnant (confirmed with positive serum pregnancy test) or breastfeeding, or planning to become pregnant.
* Female participants should refrain from breastfeeding from enrolment throughout the study and for at least 7 months after last dose of study intervention, or as dictated by local PI for SoC if longer.
* Concurrent use of systemic hormone replacement therapy or oral hormonal contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1902 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2028-11-20 (Estimated); Study Completion 2032-09-23 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) in the experimental vs control arms | Date of randomization to date of the EFS event, up to 93 months after the first subject randomized
  EFS is defined as the time from the date of randomisation until the date of the first occurrence of any of the following events: disease progression precluding surgery, disease recurrence (local, regional, distant, or contralateral), second primary invasive cancer (other than squamous or basal cell skin cancer), or relapse from prior malignancy, or death by any cause (in the absence of recurrence). Non-invasive breast cancers and positive margins in the surgical sample do not count as an event for EFS. EFS will be determined by the investigator based on all available clinical assessments.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest will be the Hazard Ratio of EFS.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) in the experimental vs control arms | At the time of definitive surgery
  pCR rate is defined as the proportion of participants who have no evidence by haematoxylin and eosin staining of residual invasive disease or lymphovascular invasion at the time of definitive surgery in the complete resected breast specimen and all sampled regional lymph nodes (ypT0/Tis ypN0) by blinded central evaluation.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest will be the difference between the pCR rates.
Overall Survival (OS) in the experimental vs control arms | Date of randomization to date of death due to any cause, up to 108 months after the first subject randomized
  Key Secondary - OS is defined as the time from the date of randomisation until the date of death due to any cause.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest will be the Hazard Ratio of OS.
Distant disease-free survival (DDFS) in the experimental vs control arms | Date of randomization to date of the DDFS event, up to 93 months after the first subject randomized
  DDFS is defined as the time from the date of randomisation until the date of the first occurrence of any of the following events: distant metastasis, occurrence of second primary invasive cancer (other than squamous or basal cell skin cancer), relapse from prior malignancy or death by any cause (in the absence of recurrence). DDFS will be determined by the investigator based on all available clinical assessments.
  The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest will be the Hazard Ratio of DDFS.
Participant-reported breast and arm symptoms in the experimental vs. control arms | From Cycle 1 Day 1 of neoadjuvant treatment until pre-surgery safety FU visit (for approximately 24 weeks) or EOT - whichever occurs first.
  Breast and arm symptoms measured by the EORTC IL116. The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest is the mean between-arm difference in breast and arm symptom scores.
Participant-reported physical function in the experimental vs. control arms | From Cycle 1 Day 1 of neoadjuvant treatment until pre-surgery safety FU visit (for approximately 24 weeks) or EOT - whichever occurs first, and then from Cycle 1 Day 1 of adjuvant treatment until EOT (for approximately 27 weeks).
  Physical function measured by the PROMIS Physical Function Short Form 8c. The analysis will include all dosed participants. The measure of interest is the mean between-arm difference in physical function scores.
Participant-reported fatigue in the experimental vs. control arms | From Cycle 1 Day 1 of neoadjuvant treatment until pre-surgery safety FU visit (for approximately 24 weeks) or EOT - whichever occurs first, and then from Cycle 1 Day 1 of adjuvant treatment until EOT (for approximately 27 weeks).
  Fatigue measured by the PROMIS Fatigue Short Form 7a. The analysis will include all dosed participants. The measure of interest will be the difference on the proportions of participants reporting different levels of fatigue and mean between-arm difference in the fatigue scores.
Participant-reported Global health status/Quality of life (GHS/QoL)in the experimental vs. control arms | From Cycle 1 Day 1 of neoadjuvant treatment until pre-surgery safety FU visit (for approximately 24 weeks) or EOT - whichever occurs first, and then from Cycle 1 Day 1 of adjuvant treatment until EOT (for approximately 27 weeks).
  Global health status/Quality of life measured by EORTC IL172. The analysis will include all randomised participants, as randomised, regardless of whether the participant withdraws from randomised therapy or receives another anticancer therapy.
  The measure of interest is the mean between-arm difference in GHS/QoL scores.
Pharmacokinetics of Dato-DXd (in combination with durvalumab) | Day 1 of cycles 1,2,4,8 (Each cycle is 21 days) and at pre-surgery safety follow up visit
  Plasma concentrations of Dato-DXd (ug/ml )
Pharmacokinetics of Dato-DXd (in combination with durvalumab) | Day 1 of cycles 1,2,4,8 (Each cycle is 21 days) and at pre-surgery safety follow up visit
  Plasma concentrations of total anti-TROP2 antibody (ug/ml )
Pharmacokinetics of Dato-DXd (in combination with durvalumab) | Day 1 of cycles 1,2,4,8 (Each cycle is 21 days) and at pre-surgery safety follow up visit
  Plasma concentrations of DXd (MAAA-1181a) (ng/ml)
Immunogenicity of Dato-DXd (in combination with durvalumab) | Day 1 of cycles 1,2,4,8 (Each cycle is 21 days) and at pre-surgery safety follow up visit
  Presence of antidrug antibodies (ADAs) for Dato-DXd (confirmatory results: positive or negative, titres).
Safety of Dato-DXd (in combination with durvalumab) | Randomization to final safety follow-up visit, either 90 days after last dose of study intervention for those who complete planned study intervention or 90 days after date of discontinuation for those who discontinue study intervention prematurely
  Safety and tolerability will be evaluated in terms of AEs graded by CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (252):
- United States (56):
  - Research Site, Daphne, Alabama
  - Research Site, Prescott, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Rogers, Arkansas
  - Research Site, Los Angeles, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Rosa, California
  - Research Site, Torrance, California
  - Research Site, Aurora, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Des Moines, Iowa
  - Research Site, Edgewood, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Annapolis, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Grand Rapids, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, Burnsville, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, East Brunswick, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Santa Fe, New Mexico
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Blue Ash, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Flower Mound, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Webster, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Tacoma, Washington
- Research Site, East Melbourne, Australia
- Austria (4):
  - Research Site, Feldkirch
  - Research Site, Innsbruck
  - Research Site, Linz
  - Research Site, Salzburg
- Belgium (6):
  - Research Site, Antwerp
  - Research Site, Brasschaat
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Libramont-Chevigny
- Brazil (11):
  - Research Site, Brasília
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Londrina
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Taubaté
  - Research Site, Vitória
- Bulgaria (2):
  - Research Site, Shumen
  - Research Site, Sofia
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Barrie, Ontario
  - Research Site, London, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Lévis, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Montreal
  - Research Site, Ottawa
- China (23):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Suining
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xintai
  - Research Site, Zhaoqing
  - Research Site, Zhengzhou
- France (13):
  - Research Site, Avignon
  - Research Site, Bayonne
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Reims
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Villejuif
- Germany (19):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Dessau
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Münster
  - Research Site, Trier
  - Research Site, Ulm
- Research Site, Hong Kong, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Szekszárd
- India (8):
  - Research Site, Bengaluru
  - Research Site, Delhi
  - Research Site, Kolkata
  - Research Site, Marg Jaipur
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, Thiruvananthapuram
  - Research Site, Vadodara
- Italy (12):
  - Research Site, Empoli
  - Research Site, Lucca
  - Research Site, Macerata
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, Torino
  - Research Site, Tricase
  - Research Site, Udine
- Japan (28):
  - Research Site, Akashi-shi
  - Research Site, Akita
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Hidaka-shi
  - Research Site, Hirakata-shi
  - Research Site, Hiroshima
  - Research Site, Isehara-shi
  - Research Site, Kashiwa
  - Research Site, Kumamoto
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Niigata
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Sunto-gun
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (4):
  - Research Site, George Town
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Selangor
  - Research Site, Kuching
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Warsaw
- Research Site, Singapore, Singapore
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seongnam
  - Research Site, Seoul
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Hospitalet deLlobregat
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Seville
  - Research Site, Zaragoza
- Switzerland (4):
  - Research Site, Baden
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Frauenfeld
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Dusit
  - Research Site, Muang
  - Research Site, Songkhla
- Turkey (Türkiye) (5):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Kayseri
  - Research Site, Samsun
- United Kingdom (7):
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Lancaster
  - Research Site, London
  - Research Site, Northampton
  - Research Site, Oxford
  - Research Site, Taunton
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hồ Chí Minh
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] McArthur HL, Tolaney SM, Dent R, Schmid P, Asselah J, Liu Q, Meisel JL, Niikura N, Park YH, Werutsky G, Bianchini G, Andersen JC, Kozarski R, Rokutanda N, Pistilli B, Loibl S. TROPION-Breast04: a randomized phase III study of neoadjuvant datopotamab deruxtecan (Dato-DXd) plus durvalumab followed by adjuvant durvalumab versus standard of care in patients with treatment-naive early-stage triple negative or HR-low/HER2- breast cancer. Ther Adv Med Oncol. 2025 Feb 5;17:17588359251316176. doi: 10.1177/17588359251316176. eCollection 2025. PMID 39917260
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/432775